CLINICAL TRIAL: NCT06596694
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of Patritumab Deruxtecan in Gastrointestinal Cancers
Brief Title: Study of Patritumab Deruxtecan in Participants With Gastrointestinal Cancers (MK-1022-011) (HERTHENA-PanTumor02)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1022-011; MK-1022-011 (Other: MSD); 2024-512442-41-00 (Registry Identifier: EU CT); U1111-1305-0677 (Registry Identifier: UTN)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patritumab deruxtecan (Experimental): Participants receive patritumab deruxtecan intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks) until disease progression, intolerable toxicity, or investigator decision.
  Interventions: Biological: Patritumab deruxtecan

INTERVENTIONS:
Biological: Patritumab deruxtecan — Administered via intravenous (IV) infusion
  Other Names: MK-1022; HER3-DXd; U3-1402

SUMMARY:
Researchers want to learn if patritumab deruxtecan (MK-1022) can treat certain gastrointestinal (GI) cancers. The GI cancers being studied are advanced (the cancer has spread to other parts of the body). The goals of this study are to learn:

* About the safety and how well people tolerate of patritumab deruxtecan
* How many people have the cancer respond (get smaller or go away) to treatment

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has one of the following cancers:

  * Unresectable or metastatic colorectal cancer.
  * Advanced and/or unresectable biliary tract cancer (BTC)
  * Hepatocellular carcinoma (HCC) not amenable to locoregional therapy
  * Locally advanced unresectable or metastatic gastroesophageal cancer
* Has received prior therapy for the cancer.
* Has recovered from any side effects due to previous cancer treatment

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of (noninfectious) interstitial lung disease (ILD) or pneumonitis that required steroids, or has current ILD or pneumonitis, and/or suspected ILD or pneumonitis that cannot be ruled out by standard diagnostic assessments at Screening
* Has clinically severe respiratory compromise (based on the investigator's assessment) resulting from intercurrent pulmonary illnesses
* Has evidence of any leptomeningeal disease
* Has clinically significant corneal disease
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2028-12-07 (Estimated); Study Completion 2028-12-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicity (DLT) (Dose-Escalation Phase) | Up to 21 days
  DLT will be defined as any drug-related adverse event observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next 21-day cycle. The number of participants in the dose-escalation phase who experience a DLT will be presented.
Number of Participants with One or More Adverse Events (AEs) | Up to approximately 44 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be presented.
Number of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 44 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Objective Response Rate (ORR) | Up to approximately 44 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 44 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression Free Survival (PFS) | Up to approximately 44 months
  PFS is defined as the time from first day of study intervention to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by BICR. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 44 months
  OS is the length of time from when the participant starts treatment until death from any cause.
Maximum Plasma Concentration (Cmax) of Patritumab Deruxtecan | At designated time points (up to ~44 months)
  Blood samples collected at protocol specific time points will be used to determine the Cmax of patritumab deruxtecan.
Trough Concentration (Ctrough) of Patritumab Deruxtecan | At designated time points (up to ~44 months)
  Blood samples collected at protocol specific time points will be used to determine the Ctrough of patritumab deruxtecan.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (62):
- United States (13):
  - UCLA Hematology Oncology Santa Monica ( Site 1205), Santa Monica, California
  - University of Colorado Cancer Center ( Site 1200), Aurora, Colorado
  - Sibley Memorial Hospital ( Site 1208), Washington D.C., District of Columbia
  - University of Florida ( Site 1202), Gainesville, Florida
  - Mount Sinai Medical Center Comprehensive Cancer Center ( Site 1213), Miami Beach, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 1203), Marietta, Georgia
  - University of Chicago Medical Center ( Site 1204), Chicago, Illinois
  - Renown Regional Medical Center ( Site 1221), Reno, Nevada
  - NYU Langone Hospital - Long Island ( Site 1230), Mineola, New York
  - Perlmutter NYU Cancer Center ( Site 1212), New York, New York
  - Scott & White Medical Center-Temple ( Site 1224), Temple, Texas
  - Oncology and Hematology Associates of Southwest Virginia (BRCC) ( Site 1207), Roanoke, Virginia
  - University of Wisconsin ( Site 1210), Madison, Wisconsin
- Australia (4):
  - Westmead Hospital ( Site 0100), Sydney, New South Wales
  - Alfred Health ( Site 0102), Melbourne, Victoria
  - Austin Health ( Site 0103), Melbourne, Victoria
  - One Clinical Research ( Site 0104), Mount Pleasant, Western Australia
- Canada (3):
  - QEII Health Sciences Centre - Victoria General Site ( Site 0200), Halifax, Nova Scotia
  - Sunnybrook Research Institute - Odette Cancer Centre ( Site 0206), Toronto, Ontario
  - McGill University Health Centre ( Site 0202), Montreal, Quebec
- Chile (4):
  - Fundacion Arturo Lopez Perez ( Site 0301), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión ( Site 0305), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 0302), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0300), Santiago, Region M. de Santiago
- China (9):
  - The First Affiliated Hospital of Anhui Medical University ( Site 0405), Hefei, Anhui
  - Fujian Provincial Cancer Hospital ( Site 0408), Fuzhou, Fujian
  - Zhongshan Hospital Fudan University (Xiamen Branch) ( Site 0412), Xiamen, Fujian
  - Southern Medical University Nanfang Hospital ( Site 0413), Fuzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University ( Site 0404), Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University ( Site 0411), Nanning, Guangxi
  - Henan Cancer Hospital ( Site 0403), Zhengzhou, Henan
  - Zhongshan Hospital,Fudan University ( Site 0400), Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University ( Site 0409), Taiyuan, Shanxi
- France (3):
  - Hopital de la Croix Rousse ( Site 0502), Lyon, Auvergne-Rhône-Alpes
  - Hopital Beaujon ( Site 0500), Clichy, Hauts-de-Seine
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 0501), Rennes, Ille-et-Vilaine
- Israel (3):
  - Rambam Health Care Campus ( Site 0603), Haifa
  - Hadassah Medical Center ( Site 0602), Jerusalem
  - Sourasky Medical Center ( Site 0601), Tel Aviv
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0700), Milan
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0701), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 0702), Roma
- Harbour Cancer & Wellness ( Site 0800), Auckland, New Zealand
- South Korea (4):
  - Seoul National University Hospital ( Site 0900), Seodaemun-gu, Seoul
  - Severance Hospital, Yonsei University Health System ( Site 0903), Seoul
  - Asan Medical Center ( Site 0902), Seoul
  - Samsung Medical Center ( Site 0901), Seoul
- Spain (4):
  - Hospital Central de Asturias ( Site 1001), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron ( Site 1000), Barcelona
  - Hospital Universitario Gregorio Maranon ( Site 1002), Madrid
  - Hospital Clinico San Carlos... ( Site 1003), Madrid
- Switzerland (2):
  - Hopitaux Universitaires de Geneve HUG. ( Site 1102), Geneva
  - Universitaetsspital Zuerich ( Site 1105), Zurich
- Taiwan (3):
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 1502), Tainan
  - National Taiwan University Hospital ( Site 1500), Taipei
  - Taipei Veterans General Hospital ( Site 1501), Taipei
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital ( Site 1301), Bangkoknoi, Bangkok
  - Ramathibodi Hospital ( Site 1302), Ratchathewi, Bangkok
- Turkey (Türkiye) (4):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi ( Site 1400), Yenimahalle, Ankara
  - Dokuz Eylul Universitesi Hastanesi ( Site 1402), Balçova, İzmir
  - Adana City Hospital ( Site 1404), Adana
  - Hacettepe Universite Hastaneleri ( Site 1401), Ankara

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26305&tenant=MT_MSD_9011